CLINICAL TRIAL: NCT04632771
Title: A Pilot Study to Evaluate the Nutritional Status of Women and Children in Northern Ghana, and Knowledge, Attitudes and Practices Related to Bouillon Cube Use
Brief Title: Nutritional Status and Bouillon Use in Northern Ghana
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: University of Ghana (Other); Newcastle University (Other); Penn State University (Other); Helen Keller International (Other)
Responsible Party: Sponsor
Other Study IDs: 1536100
Record Dates: First submitted 2020-10-27; First posted 2020-11-17 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Iron Deficiency; Vitamin A Deficiency; Vitamin B 12 Deficiency; Folate Deficiency; Zinc Deficiency; Dietary Habits; Anemia
MeSH Terms: conditions — Iron Deficiencies; Vitamin A Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Feeding Behavior; Anemia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — In the pilot survey, samples of whole blood will be collected from women of reproductive age for assessment of folate status. Samples of serum, plasma, washed red blood cells, and urine will be collected from women and children, and breast milk will be collected from lactating women. Samples will be analyzed for indicators of micronutrient status and inflammation as described in the protocol (DNA analyses will not be conducted).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Pilot survey: non-pregnant, non-lactating women: Survey of non-pregnant, non-lactating women 15-49 years of age (n=250)
  Interventions: Other: N/A (observational study)
- Pilot survey: lactating women: Survey of lactating women 15-49 years of age who are currently breastfeeding a child 4-18 months of age (n=250)
  Interventions: Other: N/A (observational study)
- Pilot survey: children: Survey of children 2-5 years of age (n=250)
  Interventions: Other: N/A (observational study)
- RID Pilot 1: Two-week study to assess total body vitamin A stores in a sample of non-pregnant, non-lactating women 15-49 years of age (n=30)
  Interventions: Other: N/A (observational study)
- RID Pilot 2: Kinetic study with "Super-woman" design to develop a prediction equation to assess total body vitamin A stores among non-pregnant, non-lactating women 15-49 years of age (n=123)
  Interventions: Other: N/A (observational study)
- Focus group discussions: Focus group discussions conducted among women of reproductive age, older women, and men (n=120 total)
  Interventions: Other: N/A (observational study)
- Market assessment: Survey of retail outlets selling fortified staple foods and/or bouillon (n=50 shop owners or operators)
  Interventions: Other: N/A (observational study)
- Recipe observations: Observations of cooking of local dishes by selected participants (n=50) enrolled in the pilot survey.
  Interventions: Other: N/A (observational study)

INTERVENTIONS:
Other: N/A (observational study) — N/A (observational study)

SUMMARY:
This pilot aims to generate data that are critical for informing the design of a planned, more detailed study to evaluate the effect of multiple micronutrient (MN)-fortified bouillon cube on biomarkers of nutrient status of women and children. Data collection includes measures of nutritional status and dietary intake among women and children and their households in communities in northern Ghana.

DETAILED DESCRIPTION:
Background: Micronutrient (MN) deficiencies are severe and widespread in West Africa including Ghana, which contributes to impaired growth and development in children, increased risk of mortality, and low economic productivity in adults. While large-scale intervention programs (including salt iodization and cooking oil and wheat flour fortification) exist, these programs are often not well-monitored, and they often provide only a subset of nutrients or reach only a subset of the deficient population.

Bouillon cubes may be an ideal fortification vehicle for delivering micronutrients in West Africa because they are purchased by most households (including rural and poorer households), added to home-made meals and consumed by most members of the household in relatively constant amounts, and they are mainly processed centrally at large scale. However, several important questions must be addressed regarding the extent to which multi-fortified bouillon cubes can address inadequate intake of key micronutrients.

Objective: This pilot aims to generate data that are critical for informing the design of a planned, more detailed study to evaluate the effect of multiple micronutrient-fortified bouillon cube on biomarkers of nutrient status of women and children.

Methods: This will be a cross-sectional study, which will be conducted in the Kumbungu and Tolon districts in the Northern Region, where a recent survey showed that micronutrient deficiencies were common. Four sets of research activities will be carried out, including:

1. Pilot survey: The investigators will recruit non-pregnant, non-lactating women of reproductive age, WRA (n = 250), children 2-5 years of age (n = 250), and lactating women (n= 250) who will be identified from households in selected communities using the random walk method. Information collected will include anthropometric and micronutrient status, hemoglobin concentration, inflammation, morbidity, household-level food consumption, and individual dietary intakes.
2. Retinol isotope dilution (RID) Pilot Study 1: The investigators will recruit non-pregnant and nonlactating women of reproductive age, WRA (n = 30) from a subset of the same communities as the pilot survey using the random walk method, and quantitatively estimate their total body vitamin A stores after consuming a dose of d6-labelled vitamin A. Total body stores of vitamin A will be estimated at 14 days after dosing.
3. Retinol isotope dilution (RID) Pilot Study 2 (kinetic study): Based on results from RID pilot study 1, the investigators will recruit non-pregnant and non-lactating women of reproductive age, WRA (n = 123) from a subset of the same communities as the pilot survey using the random walk method, to construct a population-level plasma retinol kinetic curve, after consuming a dose of d6-labelled vitamin A. A compartmental model will be fit to the plasma retinol kinetic data to develop population-specific coefficients for the RID prediction equation to quantitatively estimate total body vitamin A stores of WRA in the study population.
4. Formative research: The investigators will (a) conduct focus group discussions on knowledge, attitudes and practices related to salt and bouillon cube use, nutrition and health problems in the community, and micronutrient fortification; (b) perform a market assessment of the availability and cost of fortified, non-fortified and potentially fortifiable foods in the communities; and (c) observe how various local food recipes are prepared, including the types and quantities of ingredients used, and cooking duration and temperature.

ELIGIBILITY:
Pilot survey

Inclusion Criteria:

* non-pregnant, non-lactating woman of reproductive age (15-49 years) OR child 2-5 years of age OR non-pregnant lactating woman (4-18 mo post-partum, 15-49 years of age)
* signed informed consent by participant (if adult woman) or by at least one parent or guardian (if child)

Exclusion Criteria:

* severe illness warranting hospital referral
* chronic severe medical condition (e.g. malignancy) or congenital anomalies requiring frequent medical attention or potentially inferring with nutritional status
* unable to provide informed consent due to impaired decision making abilities (if adult woman, or caretaker of potentially eligible child)
* current participation in a clinical trial

RID Pilot 1

Inclusion Criteria:

* non-pregnant, nonlactating woman of reproductive age (15-49 years)
* signed informed consent
* planning to remain in the study area for the next 1 month
* not planning to become pregnant during the next 1 month

Exclusion Criteria:

* unable to provide informed consent due to impaired decision making abilities
* pregnancy (as ascertained via urine pregnancy test for human chorionic gonadotropin)
* severe illness warranting hospital referral
* reported fever, vomiting or diarrhea (> 3 liquid or semi-liquid stools in 24h) in 7 d prior to data collection
* chronic medical condition (e.g. malignancy, gastrointestinal disease) or congenital anomalies requiring frequent medical attention or potentially inferring with nutritional status
* current participation in a clinical trial
* hemoglobin concentration <80 g/L on the day of isotope dosing
* C-reactive protein concentration > 5 mg/L on the day of isotope dosing
* reported use of micronutrient supplements that contain vitamin A more than 1 time/wk in the past 30 days

RID Pilot 2

Inclusion Criteria:

* non-pregnant, nonlactating woman of reproductive age (15-49 years)
* signed informed consent
* planning to remain in the study area for the next 4 months
* not planning to become pregnant during the next 4 months

Exclusion Criteria:

* unable to provide informed consent due to impaired decision making abilities
* pregnancy (as ascertained via urine pregnancy test for human chorionic gonadotropin)
* severe illness warranting hospital referral
* reported fever, vomiting or diarrhea (> 3 liquid or semi-liquid stools in 24h) in 7 d prior to data collection
* chronic medical condition (e.g. malignancy, gastrointestinal disease) or congenital anomalies requiring frequent medical attention or potentially inferring with nutritional status
* current participation in a clinical trial
* hemoglobin concentration <80 g/L on the day of isotope dosing
* C-reactive protein concentration > 5 mg/L on the day of isotope dosing
* reported use of micronutrient supplements that contain vitamin A more than 1 time/wk in the past 30 days

Formative Research

Inclusion Criteria:

* Adults (including women, men, and other key community members such as merchants, etc.)
* Provision of written informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Households in the urban and rural areas in Tolon and Kumbungu districts, in northern Ghana
Sampling Method: Non-Probability Sample
Enrollment: 995 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | Day 1
  Hemoglobin concentration in venous blood (g/dL) among women and children
Iron status | Day 1
  Concentrations of iron status biomarkers (serum iron, ferritin, and soluble transferrin receptor) among women and children
Vitamin A status | Day 1
  Concentrations of vitamin A status biomarkers (serum retinol and retinol-binding protein) among women and children
Vitamin B12 status | Day 1
  Concentrations of vitamin B12 in serum among women and children
Folate status | Day 1
  Concentrations of folate in serum (among women and children) and whole blood and erythrocytes (women only)
Zinc status | Day 1
  Serum zinc concentration among women and children
Breast milk vitamin A concentration | Day 1
  Vitamin A concentration in breast milk, expressed per unit volume and per gram fat
Breast milk vitamin B12 concentration | Day 1
  Vitamin B12 concentration in breast milk
Total body vitamin A stores | Day 7
  Distribution of total body vitamin A stores among non-pregnant, non-lactating women, expressed as total mass and per gram of liver, estimated by retinol isotope dilution
Total body vitamin A stores | Day 14
  Distribution of total body vitamin A stores among non-pregnant, non-lactating women, expressed as total mass and per gram of liver, estimated by retinol isotope dilution
Coefficient "Fa" | Blood samples from RID Pilot 2 participants collected at randomly assigned time points over a 90-day time frame
  Defined as the fraction of the oral tracer dose absorbed and retained in stores, estimated by modeling of data on labeled and unlabelled vitamin A in plasma collected using a "Super Woman" design and used to calculate total body stores for individual participants.
Coefficient "S" | Blood samples from RID Pilot 2 participants collected at randomly assigned time points over a 90-day time frame
  Defined as retinol specific activity in plasma/stores at time "t", estimated by modeling of data on labeled and unlabelled vitamin A in plasma collected using a "Super Woman" design and used to calculate total body stores for individual participants.
Prevalence of anemia and micronutrient deficiencies | Day 1
  Prevalence of hemoglobin and micronutrient biomarkers above or below relevant cutoffs
Urinary iodine concentration | Day 1
  Iodine concentration of urine among women and children
Themes from focus group discussions | Day 1
  Perceptions of bouillon and salt use, cooking practices, noncommunicable disease, and other nutrition and diet-related issues
Recipe ingredients | Day 1
  Quantity of each recipe ingredient (including bouillon and salt) used in common local recipes; interpreted in relation to cooking duration and temperature (type and duration, e.g. of boiling) used in common recipes
Fortified food accessibility | Day 1
  Availability, price, and fortification levels of fortified food products in markets

SECONDARY OUTCOMES:
Blood pressure | Day 1
  Blood pressure measured among women and children (mm Hg, systolic and diastolic)
Hypertension | Day 1
  Prevalence of blood pressure measurements above cutoffs for hypertension
Height, cm | Day 1
  Standing height measured among women and children
Weight, kg | Day 1
  Weight measurement among women and children
Waist to hip ratio | Day 1
  Waist and hip circumference (measured in cm) among women and their ratio
Mid-upper arm circumference, cm | Day 1
  Mid-upper arm circumference measured among children
Anthropometric Z-scores | Day 1
  Z-scores calculated for young children based on WHO growth standards (height-for-age, weight-for-height, height-for-age, BMI-for-age)
Prevalence of undernutrition | Day 1
  Prevalence of anthropometric Z-scores or mid-upper arm circumference below WHO cutoffs to indicate child undernutrition
Prevalence of overweight and obesity | Day 1
  Prevalence of body mass index (women) or BMI-for-age Z-score (children) above WHO cutoffs
Morbidity symptoms | Day 1
  Reported malaria, diarrhea, fever, or vomiting in the past 7 days (all survey participants)
Inflammation | Day 1
  Serum concentrations of CRP, AGP, amyloid A, MCP-1, IL-6, IL-10, IL-1b, adiponectin
Household-food consumption | Day 1
  Calculated daily household level consumption and individual apparent consumption of fortified foods (wheat flour, oil, salt) and bouillon estimated using 1-month recall
Individual dietary intake | Day 1
  Dietary intake of fortified foods and bouillon, measured by 24h recall among a subset of women participating in the survey who also participate in cooking observations
Urinary sodium concentration | Day 1
  Expressed per unit volume and in relation to urinary creatinine concentration
Status of other micronutrients | Day 1
  Concentrations of micronutrients in serum and breast milk (vitamins E, B1, B2, B3, B5, B6, B7)

OTHER OUTCOMES:
Micronutrient supplement use | Day 1
  Reported use of daily or periodic micronutrient supplements in the past month
Consumption of fruits and vegetables | Day 1
  Assessed using the WHO STEPS questionnaire
Consumption of snacks and sweetened beverages | Day 1
  Assessed using the WHO STEPS questionnaire
Physical activity | Day 1
  Assessed using the WHO STEPS questionnaire
Tobacco use | Day 1
  Assessed using the WHO STEPS questionnaire
Alcohol use | Day 1
  Assessed using the WHO STEPS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Green MH, Lopez-Teros V, Green JB, Lietz G, Kumordzie SM, Oxley A, Fuseini AD, Nyaaba KW, Becher E, Davis JN, Wessells KR, Adu-Afarwuah S, Engle-Stone R, Haskell MJ. Use of Population-Based Compartmental Modeling and Retinol Isotope Dilution to Study Vitamin A Kinetics and Total Body Stores among Ghanaian Women of Reproductive Age. Curr Dev Nutr. 2024 Oct 18;8(11):104484. doi: 10.1016/j.cdnut.2024.104484. eCollection 2024 Nov. PMID 39634788
- [Derived] Davis JN, Kumordzie SM, Arnold CD, Wessells KR, Nyaaba KW, Adams KP, Tan XJ, Becher E, Vosti SA, Adu-Afarwuah S, Engle-Stone R. Consumption of Discretionary Salt and Salt from Bouillon among Households, Women, and Young Children in Northern Region, Ghana: A Mixed-Methods Study with the Condiment Micronutrient Innovation Trial (CoMIT) Project. Curr Dev Nutr. 2024 Feb 6;8(3):102088. doi: 10.1016/j.cdnut.2024.102088. eCollection 2024 Mar. PMID 38419834